CLINICAL TRIAL: NCT02904564
Title: Conventional Microneedling Compared to Microneedling Associated With 5-FU Infusion (Microinfusion of Medication Into the Skin - MMP) for Idiopathic Guttate Hypomelanosis (IGH) Repigmentation
Brief Title: Conventional Microneedling vs Microneedling With 5-FU (MMP) for Idiopathic Guttate Hypomelanosis (IGH) Repigmentation
Acronym: MMP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Dermatologica Arbache ltda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2016-08-26; First posted 2016-09-19 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Photosensitivity Disorders
Keywords: drug delivery; Idiopathic Guttate Hypomelanosis
MeSH Terms: conditions — Photosensitivity Disorders | interventions — Matrix Metalloproteinases; Fluorouracil; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMP with 5-FU infusion (Experimental): MMP with 5-FU infusion using tattoo device
  Interventions: Drug: MMP with 5-FU
- MMP with saline infusion (Placebo Comparator): MMP with saline infusion using tattoo device
  Interventions: Drug: MMP with Saline infusion

INTERVENTIONS:
Drug: MMP with 5-FU — MMP with 5-FU using tattoo device
  Other Names: 5-fluorouracil; drug delivery; drug infusion; microinfusion of medication percutaneously; MMP
  Arms: MMP with 5-FU infusion
Drug: MMP with Saline infusion — MMP with saline infusion using tattoo device
  Other Names: MMP
  Arms: MMP with saline infusion

SUMMARY:
The purpose of this study is to determine whether 5-FU infusion (Microinfusion of Medicine Percutaneously - MMP) is effective for Idiopathic Guttate Hypomelanosis (IGH) repigmentation compared to conventional Microneedling. MMP is a procedure done with tattoo devices using medication in place of ink.

DETAILED DESCRIPTION:
Split body design. Each upper limb will receive a different intervention (experimental or placebo)

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, between ages 30 and 70
* Photodamaged skin on upper limbs with IGH lesions meeting aforementioned criteria and excluding differential diagnosis
* Fitzpatrick skin types III - V
* Apt and willing to comply with the entire program as well as appointments, treatment and examination
* Capable of understanding and providing a written informed consent
* Fertile women will have to use a viable birth control method for at least 3 months prior to entry and throughout the entire study

Exclusion Criteria:

* Pregnancy, intention to become pregnant during the course of the study, less than 3 months after delivery or less than 6 weeks after breastfeeding cessation.
* Uncontrolled comorbidity or any disease that, in the investigator's opinion, may interfere with the treatment, healing or cure.
* Present symptoms of hormonal disturbances, as per the investigator's criteria.
* Constitutional photosensitivity or due to metabolic disfunction, or due to use of external agentes (pharmaco, natural products, etc.) prior to initial treatment or during the study.
* Use of oral isotretinoin 6 months prior to initial treatment or during the course of the study.
* Prior treatment in target área 3 months prior to initial treatment or during the course of the study.
* Adverse reaction to any external agentes (gel, lotions or anesthetic creams) required during the study in case no alternative is available for such agent.
* History of keloids or other type of hypertrophic scar formation or poor wound healing in a previously injured area of skin.
* History of collagen disease.
* Displastic nevus or suspicious carcinogenic lesion in área to be treated.
* Hemmorragic disorder or under anticoagulant medication, including the use of aspirin not permitting a minimum 10-day suspension prior to each treatment period (in accordance with the criteria of the patient's physician).
* Skin frailty of sensitivity, favoring hemmorrage.
* History of immunosuppresion / immunological deficiency disorders (including HIV infection) or use of immunosuppressant medication.
* Participation in a study involving medication or another device three months prior to the study or during enrollment herein.
* Any condition which, in the investigator's opinion, would jeopardize the study or its participants, such as acute psychiatric disorders, panic syndrome or any aversion to needles or to the procedure.
* Hypochromiant dermatoses such as vitiligo, pitiriasis, versicolor, albinism.
* Dermatoses that evolve like Koebner's phenomenon.
* Cutaneous infectious process at the application site.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-20 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Lesions counting of Idiopathic Guttate Hypomelanosis (IGH) | 30 days
  Two assessors will independently count the number of lesions in the treated skin area

SECONDARY OUTCOMES:
Patient satisfaction assessed by Likert scale | 30 days
  self-administered
Local adverse events | 30 days
  Frequency of patients presenting at least one local adverse event (ex:intense pain, scars, infection)
Systemic adverse events | 24 hours
  Frequency of patients presenting at least one systemic adverse event (anaphylactic reaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dermatologica Arbache Ltda, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arbache S, Hirata SH. Efficacy and Safety of 5-Fluorouracil Tattooing to Repigment Idiopathic Guttate Hypomelanosis: A Split-Body Randomized Trial. Dermatol Surg. 2023 Jun 1;49(6):603-608. doi: 10.1097/DSS.0000000000003793. Epub 2023 Apr 3. PMID 37011024